CLINICAL TRIAL: NCT06928129
Title: Clinical Feasibility of the BinaxNOW™ COVID-19/Flu A&B Combo in the Southern Hemisphere
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2506401
Record Dates: First submitted 2025-04-10; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Influenza Type A; Influenza Type B; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Study staff will collect two (2) anterior nasal swabs from each Participant.
  The Participant will self-collect one (1) anterior nasal swab, perform the BinaxNOW™ COVID-19/Flu A&B Combo, then interpret and record the result.
  Site staff will collect one (1) anterior nasal swab from the Participant by inserting the swab up to 1 inch into one of the anterior naris. Staff will rotate the swab against the nasal mucosa five (5) times to obtain sample and withdraw. Staff will repeat with the other anterior naris using the same swab, and vigorously elute the swab in Viral Transport Medium (VTM)/Universal Transport Media (UTM) immediately (within 5 minutes) of sample collection. The swab should be rotated vigorously in the VTM/UTM liquid for 10 seconds. The swab head will be left in the VTM/UTM, by snapping the shaft or clipping the base of the swab if necessary
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Experimental: Nasal sampling/Testing (Self-Test) (Experimental): Each Participant will be provided a single-use test kit containing a BinaxNOW™ COVID-19/Flu A&B Combo, buffer and a sterile nasal swab. The Participant will self-collect one (1) anterior nasal swab, perform the BinaxNOW™ COVID-19/Flu A&B Combo, then interpret and record the result. The testing will be completed in a home like setting. After the anterior nasal swab is collected, the operator or delegated study staff will collect one anterior nasal swab from both nostrils of the subject for RT-PCR testing. VTM samples will be shipped daily to the central lab for testing with the RT-PCR protocols for Flu A, Flu B and SARS-CoV-2.
  The order of collections will be based off the subject number.
  Interventions: Diagnostic Test: BinaxNOW™ COVID-19/Flu A&B Combo Self-Test

INTERVENTIONS:
Diagnostic Test: BinaxNOW™ COVID-19/Flu A&B Combo Self-Test — Diagnostic Test: BinaxNOW™ COVID-19/Flu A&B Combo Self-Test
  The BinaxNOW™ COVID-19/Flu A&B Combo Self-Test is a visually read lateral flow in vitro immunoassay for the qualitative detection and differentiation of the nucleocapsid protein antigen to SARS-CoV-2, Influenza A, and Influenza B directly in anterior nasal swab specimens from individuals with signs and symptoms of respiratory infection.

SUMMARY:
The study is designed as a clinical feasibility, to investigate the positive and negative percent agreement (PPA and NPA) of the BinaxNOW™ COVID-19/Flu A&B Combo against a highly sensitive PCR method(s) in symptomatic patients suspected of SARS-CoV-2 or influenza infection when nasal swabs are self-collected by the patient/lay user.

DETAILED DESCRIPTION:
Approximately 700 symptomatic participants will be enrolled to achieve at least 61 COVID PCR positive, 45 Flu A PCR positives, 30 Flu B PCR positives and 301 COVID and Influenza PCR negatives.

The total number of research-related anterior nasal swabs collected from each consented Participant is two (2). Participants ages two (2) years and older meeting eligibility criteria will be enrolled.

The order of nasal swab collection will be randomized according to the Participant ID as to which swab is used for BinaxNOW™ COVID-19/Flu A&B Combo and which is to be eluted into VTM/UTM and will have the swab head left in the media (snap off or clip shaft) for comparator testing.

For Participants with an odd numbered Participant ID, the first swab will be self-collected and used for the BinaxNOW™ COVID-19/Flu A&B Combo. The second swab will be collected by a healthcare professional and eluted into VTM/UTM and will have the swab head left in the media (snap off or clip shaft) for comparator testing. The Participant will review the Instructions for Use, collect the nasal swab, and perform the BinaxNOW™ COVID-19/Flu A&B Combo, then interpret and record the result at the time specified in the product instructions.

For Participants with an even numbered Participant ID, the first swab will be collected by a healthcare professional and eluted into VTM/UTM and will have the swab head left in the media (snap off or clip shaft) for comparator testing. The second swab will be self-collected and used for the BinaxNOW™ COVID-19/Flu A&B Combo. Once the healthcare provider collected the swab for the comparator test the Participant will review the Instructions for Use.

The VTM/UTM samples will be stored, handled, and tested with comparator assays according to the manufacturers' product instructions. VTM/UTM specimens can be stored for up to 48 hours at 2-8°C. If delivery and processing of samples exceeds specified time periods, specimens should be transported in dry ice and once in laboratory frozen at -70°C or colder.

Each Participant's demographic data, inclusion/exclusion data, days of symptom onset, comparator results, Education level, occupation, and socioeconomic status and other data points will be documented on the data collection worksheets and EDC.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least two (2) years of age, AND Participant is suspected of acute viral respiratory infection by a healthcare professional, AND
* Participant is within five (5) days of symptom onset, AND

Participant is experiencing two or more of the following symptoms:

Fever of >100.0°F/ 37.8°C or chills, Cough, Fatigue, New loss of taste or smell, Congestion or runny nose, Shortness of breath or difficulty breathing, Sore throat, Muscle or body aches, Headache

-The Participant and/or legally authorized representative is willing to undergo the informed consent/Assent process prior to study participation. A minor will need the documented consent of their parent or legal guardian unless the site has an HREC waiver for parental consent for minors.

Exclusion Criteria:

* Participant is currently enrolled in a study to evaluate an investigational drug or experimental treatment
* Participants with an active nosebleed
* Participant has undergone a nasal wash or nasal aspirate procedure on day of enrolment
* Participant has tested positive for COVID-19 within the last 45 days
* Participant has received a nasal vaccine (i.e. FluMist®) within the past 30 days.
* Participant has received antiviral medications for Influenza (Amantadine, Rimantadine, Ribavirin, Oseltamivir, Zanamivir) in the previous 45 days.
* Participant has received medication or treatment for COVID-19 infection in the last 45 days (including antivirals (such as Paxlovid), convalescent plasma therapy, monoclonal antibody treatment (mAb), Remdesivir, long-acting antibody (LAAB) treatment (Evusheld)
* Participant is unable to meet all inclusion criteria as listed above

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the positive percent agreement (PPA) and negative percent agreement (NPA) | 5 months
  The primary objective of this study is to demonstrate the positive and negative percent agreement (PPA and NPA) of the BinaxNOW™ COVID-19/Flu A&B Combo against a highly sensitive PCR method(s) in symptomatic patients suspected of SARS-CoV-2 or influenza infection when nasal swabs are self-collected by the patient/lay user. The patient/lay user will perform the test, read, and interpret the test result.

SECONDARY OUTCOMES:
Demonstrate the accuracy of the BinaxNOW™ COVID-19/Flu A&B Combo Self-Test in patient/lay user | 5 months
  The secondary objective of this study is to demonstrate the accuracy of the BinaxNOW™ COVID-19/Flu A&B Combo Self-Test in the hands of patients/lay users, which are "intended users" in a point of care (POC) Clinical Laboratory Improvement Amendments of 1988 (CLIA) moderate, high or waived complexity test environment

IPD SHARING:
Plan to Share IPD: No
No plans to share as this is a feasibility trial.